CLINICAL TRIAL: NCT06221787
Title: Stem Cell Derived Exosomes in the Treatment of Melasma and Its Percutaneous Penetration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, ChenXiaosong, Director of Plastic Surgery and Regenerative Medicine, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020KY0155
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Melasma
Keywords: Melasma; Stem cell-derived exosomes; Percutaneous Penetration
MeSH Terms: conditions — Melanosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1565 nm non-ablative fractional laser combined with normal saline (Placebo Comparator): The treatment parameters were adjusted according to each patient's age, skin color, surface area of affected skin, location of melasma, and skin type.After the scanning, infusing with normal saline in the entire face.
  Interventions: Procedure: 1565 nm non-ablative fractional laser combined with normal saline
- microneedles combined with hUCMSC-Exos (Experimental): The hUCMSC-Exos were applied while rolling a microneedle roller in the entire face.
  Interventions: Procedure: microneedles combined with hUCMSC-Exos
- 1565 nm non-ablative fractional laser combined with hUCMSC-Exos (Experimental): The treatment parameters were adjusted according to each patient's age, skin color, surface area of affected skin, location of melasma, and skin type.After the scanning, infusing with hUCMSC-Exos in the entire face.
  Interventions: Procedure: 1565 nm non-ablative fractional laser combined with hUCMSC-Exos
- PBASM combined with hUCMSC-Exos (Experimental): 4-5 levels of intensity were used, rolling each area for 8-10 min before applying the hUCMSC-Exos in the entire face.
  Interventions: Procedure: PBASM combined with hUCMSC-Exos

INTERVENTIONS:
Procedure: 1565 nm non-ablative fractional laser combined with normal saline — After 1565 nm non-ablative fractional laser treatment, patients with melasma were smeared with normal saline and to compared with those smeared with exosomes after laser treatment.
  Arms: 1565 nm non-ablative fractional laser combined with normal saline
Procedure: microneedles combined with hUCMSC-Exos — the hUCMSC-Exos were applied while rolling a microneedle roller and to compared with those used 1565 nm non-ablative fractional laser or PBASM combined with hUCMSC-Exos.
  Arms: microneedles combined with hUCMSC-Exos
Procedure: 1565 nm non-ablative fractional laser combined with hUCMSC-Exos — After 1565 nm non-ablative fractional laser treatment, patients with melasma were smeared with hUCMSC-Exos and to compared with those smeared with normal saline after laser treatment.What's more,compared with those used microneedles or PBASM combined with hUCMSC-Exos.
  Arms: 1565 nm non-ablative fractional laser combined with hUCMSC-Exos
Procedure: PBASM combined with hUCMSC-Exos — a plasma named Peninsula Blue Aurora Shumin Master (PBASM) rolling each area for 8-10 min before applying the hUCMSC-Exos in the entire face. And to compared with those used 1565 nm non-ablative fractional laser or microneedles combined with hUCMSC-Exos.
  Arms: PBASM combined with hUCMSC-Exos

SUMMARY:
Melasma is a refractory skin disease due to its complex pathogenesis and difficult treatment. Studies have found that human umbilical cord mesenchymal stem cell-derived exosomes (hUCMSC-Exos) could serve as a novel cell-free therapeutic strategy in regenerative and aesthetic medicine. It could potentially treat melasma, but the skin barrier is a challenge. This study aims to explore the safety and efficacy of hUCMSC-Exos in the treatment of melasma and means to promote its percutaneous penetration.

DETAILED DESCRIPTION:
80 patients with melasma treated in our department were divided into four groups. 1565 nm nonablative fractional laser (NAFL) combined with normal saline treatment group was used for Group A. Microneedle，NAFL，a plasma named Peninsula Blue Aurora Shumin Master (PBASM) combined with hUCMSC-Exos were used for the other treatment groups (B, C, and D, respectively). The treatment was given four times with an interval of one month. The degree of pain post-treatment, MASI, improvement rate, physician global assessment score, satisfaction and complications after treatment were evaluated six months later.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with chloasma who meet the clinical diagnostic standards and efficacy standards (revised version) of chloasma and have skin lesions on the face.

It is hoped that exosomes combined with 1565 non-ablative fractional laser, blue aurora or micro-needle can improve facial chloasma.

Fully understand and understand the content and significance of this study, implementation plan, possible benefits, risks and countermeasures, rights and obligations of subjects (including privacy protection, free withdrawal), willing to participate in this clinical study and able to cooperate well, Those who signed the informed consent form.

Exclude post-inflammatory pigmentation, malar brown-green nevus, Riehl's melanosis, pigmented lichen planus and other skin diseases.

Subjects who agree not to use other cosmetic treatments related to the study during the study period.

Exclusion Criteria:

1. Patients who refuse to sign the informed consent form to participate in the trial;
2. Those with a history of important organ diseases, or a history of autoimmune diseases or immune dysfunction;
3. Abnormal coagulation function, current use of anticoagulants, thrombophilia and history of familial genetic diseases;
4. Pregnant or lactating women;
5. Patients taking oral contraceptives or hormone replacement therapy during the study period or within the past 12 months;
6. Patients with scar constitution;
7. Active skin infection;
8. Those who have a history of multiple severe allergies, a history of hereditary allergies, photosensitivity or photosensitivity drugs, such as sulfa drugs and tetracyclines, those who are allergic to local anesthetics and those who are allergic to lidocaine components, and those who plan to undergo detoxification during the study Allergy healer;
9. History of post-inflammatory pigmentation;
10. Those who have received treatment for chloasma in the past;
11. Those who have undergone chemical peeling, dermabrasion or other skin resurfacing on their face in the past;
12. Patients who are participating in other clinical studies;
13. Other reasons that the researcher considers unsuitable for clinical investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
melasma area and severity index （MASI） | 6 months
  MASI=0.3(DMR+HMR)AMR+0.3(DF+HF)AF+0.3(DML+HML)AML+0.1(DC+HC)AC, A is the area proportion of chloasma, D is the color depth of the spots, H is the color uniformity, F is the forehead; ML is the left cheek; MR is the right cheek; C is the mandible. Scores for color depth and color uniformity of stains: total score is 4 points each, and the color degree of stains is 0 (no deepening), 1 (slightly deepened), 2 (moderately deepened), 3 (obviously deepened), 4 points (severely deepened); color uniformity is 0 points (extremely inconsistent), 1 point (slightly consistent), 2 points (moderately consistent), 3 points (obviously consistent), 4 points (almost completely consistent); damage Area proportion score: total score is 6 points, 0 is normal, 1 is <10%, 2 is 10%~29%, 3 is 30%~49%, 4 is 50%~69%, 5 It is divided into 70% to 89% and 6 points to 90% to 100%. The total score is 48 points, and the lower the score, the less serious the chloasma.

CONTACTS AND LOCATIONS:
Overall Officials: xiaosong chen, director, Study Chair — Affiliated Union Hospital of Fujian Medical University
Locations (1):
- Affiliated Union Hospital of Fujian Medical University, Fuzhou, Fujian, China